CLINICAL TRIAL: NCT02252263
Title: A Phase I Open Label Dose Escalation and Randomized Cohort Expansion Study of the Safety and Tolerability of Elotuzumab (BMS-901608) Administered in Combination With Either Lirilumab (BMS-986015) or Urelumab (BMS-663513) in Subjects With Multiple Myeloma
Brief Title: A Phase I Open Label Study of the Safety and Tolerability of Elotuzumab (BMS-901608) Administered in Combination With Either Lirilumab (BMS-986015) or Urelumab (BMS-663513) in Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA223-028
Record Dates: First submitted 2014-09-26; First posted 2014-09-30 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; lirilumab; urelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Elotuzumab + Lirilumab (Experimental): Elotuzumab weekly for 8 wks and every 2 wks thereafter + Lirilumab every 4 wks Intravenous solution for Up to 2 yrs, depending on response
  Interventions: Drug: Elotuzumab; Drug: Lirilumab
- Arm 2: Elotuzumab + Urelumab (Experimental): Elotuzumab weekly for 8 wks and every 2 wks thereafter + Urelumab every 4 wks Intravenous solution for Up to 26 weeks, depending on response
  Interventions: Drug: Elotuzumab; Drug: Urelumab

INTERVENTIONS:
Drug: Elotuzumab
  Other Names: BMS-901608
Drug: Lirilumab
  Other Names: BMS-986015
  Arms: Arm 1: Elotuzumab + Lirilumab
Drug: Urelumab
  Other Names: BMS-663513
  Arms: Arm 2: Elotuzumab + Urelumab

SUMMARY:
To assess the safety and tolerability, characterize the dose limiting toxicities (DLTs) and identify the maximally tolerated dose (MTD) of Elotuzumab administered in combination with either Lirilumab or Urelumab in subjects with multiple myeloma.

DETAILED DESCRIPTION:
Allocation:

* Part1: Non-randomized
* Part2: Randomized

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects must have histological confirmation of multiple myeloma with measurable disease (per International Myeloma Working Group (IMWG) criteria):

  * Relapsed/refractory multiple myeloma, subjects who are post autologous transplant and have achieved very good partial response (VGPR) or complete response (nCR) with minimal residual disease (MRD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Safety as measured by the rate of AEs, SAEs, deaths is the primary endpoint of this Phase 1 study. All subjects who receive at least one (full or partial) dose of Elotuzumab, Lirilumab or Urelumab will be evaluated for safety | During treatment and first 100 days after treatment
  adverse events (AEs), serious adverse events (SAEs)

SECONDARY OUTCOMES:
Best Overall Response (BOR) | At different timepoints approximately up to 2.5 years
Objective Response rate (ORR) | At different timepoints approximately up to 2.5 years
Median Duration of Response (mDOR) | At different timepoints approximately up to 2.5 years
Median Time to Response (mTTR) | At different timepoints approximately up to 2.5 years
Progression-free survival rate (PFSR) | At different timepoints approximately up to 2.5 years
M-protein levels | At different timepoints approximately up to 2.5 years
Minimal Residual Disease (MRD) status for Post Autologous Transplant subjects | At different timepoints approximately up to 2.5 years
Maximum concentration of Urelumab (Cmax) | At different timepoints approximately up to 2.5 years
Maximum concentration of Lirilumab (Cmax) | At different timepoints approximately up to 2.5 years
Area under the Curve (AUCTAU) of Urelumab | At different timepoints approximately up to 2.5 years
Area under the Curve (AUCTAU) of Lirilumab | At different timepoints approximately up to 2.5 years
Volume of distribution (Vz) for Urelumab | At different timepoints approximately up to 2.5 years
Total Clearance (CLT) of Urelumab | At different timepoints approximately up to 2.5 years
Total Clearance (CLT) of Lirilumab | At different timepoints approximately up to 2.5 years
Concentration at the end of infusion (ceoinf) of Urelumab | At different timepoints approximately up to 2.5 years
Concentration at the end of infusion (ceoinf) of Elotuzumab | At different timepoints approximately up to 2.5 years
Concentration at the end of infusion (ceoinf) of Lirilumab | At different timepoints approximately up to 2.5 years
Cmin will be capture at steady state of all study subjects | At different timepoints approximately up to 2.5 years
Occurence of Specific anti-drug antibodies (ADA) to each study drug | At different timepoints approximately up to 2.5 years
ADA status of the subject Biomarkers: NK and T cell numbers, Phenotypic and functional measures in cohort expansion subjects | At different timepoints approximately up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (6):
  - University Of Arkansas For Medical Sciences, Little Rock, Arkansas
  - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University Of Pennsylvania, Philadelphia, Pennsylvania
- Local Institution, Pamplona, Navarre, Spain

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx